CLINICAL TRIAL: NCT05696457
Title: Effects of Music Therapy in Controlling Symptoms in Patients With Acute Myeloblastic Leukemia and Undergoing Hematopoietic Stem Cell Transplantation: a Randomized Controlled Clinical Trial
Brief Title: Effects of Music Therapy in Controlling Symptoms in Patients With AML and Undergoing HSCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EC086-20
Record Dates: First submitted 2022-11-24; First posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Acute Myeloblastic Leukemia; Hematopoietic Stem Cell Transplantation
Keywords: Acute Myeloblastic Leukemia; Hematopoietic Stem Cell Transplantation; Music therapy; Symptom control
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- AML-E (Experimental): Acute myeloblastic leukemia - experimental
  Interventions: Behavioral: Passive music therapy
- AML-C (No Intervention): Acute myeloblastic leukemia - control
- AlloSCT-E (Experimental): Allogeneic stem cell transplantation - experimental
  Interventions: Behavioral: Passive music therapy
- AlloSCT-C (No Intervention): Allogeneic stem cell transplantation - control
- AutoSCT-E(I) (Experimental): Autologous stem cell transplantation - experimental (inpatient)
  Interventions: Behavioral: Passive music therapy
- AutoSCT-C(I) (No Intervention): Autologous stem cell transplantation - control (inpatient)
- AutoSCT-E(O) (Experimental): Autologous stem cell transplantation - experimental (outpatient)
  Interventions: Behavioral: Passive music therapy
- AutoSCT-C(O) (No Intervention): Autologous stem cell transplantation - control (outpatient)

INTERVENTIONS:
Behavioral: Passive music therapy — Patients included in the experimental group receive a 25 min passive music therapy session on a daily basis, which changes depending on their emotion.
  Arms: AML-E; AlloSCT-E; AutoSCT-E(I); AutoSCT-E(O)

SUMMARY:
The goal of this clinical trial is to test passive music therapy in patients receiving induction chemotherapy for an acute myeloblastic leukemia or undergoing an hematopoietic stem cell transplantation. The main questions it aims to answer are:

- Can music therapy control physical and psychological symptoms and improve the mood and quality of life of these patients?

Participants will be randomly assigned to the control and experimental group. Patients included in both groups will complete weekly mood and quality of life questionnaires. Those included in the experimental group will also complete daily symptom burden questionnaires before and after listening to a music therapy session.

Researchers will confirm if the experimental group improves their symptoms after the music therapy session and will compare both groups to see if there are differences in mood and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old.
* Patients receiving induction chemotherapy for a newly diagnosed acute myeloblastic leukemia (except for acute promyelocytic leukemia).
* Patients undergoing autologous or allogeneic stem cell transplantation.
* Being able to understand and read Spanish properly.
* Basic computer skills.

Exclusion Criteria:

* Moderate-severe hearing impairment (unilateral or bilateral).
* Past history of psychiatric disorders.
* Performance status: ECOG ≥ 3.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2022-11-21 (Actual)

PRIMARY OUTCOMES:
Change in physical and psychological symptom burden | The ESAS global score is measured before and after the daily music therapy session (from date of randomization until the date of discharge, up to 8 weeks)
  Edmonton Symptom Assessment System (ESAS) global score (0 to 110 points, higher scores mean higher symptom burden)

SECONDARY OUTCOMES:
Anxiety and depression assessed by the Hospital Anxiety and Depression Scale (HADS) score | Once a week (from date of randomization until the date of discharge, up to 8 weeks)
  HADS score (0 to 42 points, higher scores mean higher anxiety/depression)
Quality of life assessed by the Functional Assessment of Cancer Therapy - General (FACT-G) score | Once a week (from date of randomization until the date of discharge, up to 8 weeks)
  FACT-G score (0 to 108 points, higher scores mean better quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Lázaro García, MD, Principal Investigator — Fundación Jiménez Díaz University Hospital
Locations (1):
- Instituto Investigacion Sanitaria Fundacion Jimenez Diaz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lazaro-Garcia A, Lainez-Gonzalez D, Gonzalez-Rodriguez M, Cano Alsua S, Suarez M EU, Solan-Blanco L, Cornago-Navascues J, Lopez-Lorenzo JL, Llamas-Sillero P, Alonso-Dominguez JM. Music Listening in Stem Cell Transplantation and Acute Myeloid Leukemia: A Randomized Clinical Trial. J Pain Symptom Manage. 2024 Jun;67(6):501-511.e12. doi: 10.1016/j.jpainsymman.2024.02.567. Epub 2024 Mar 4. PMID 38447622